CLINICAL TRIAL: NCT07123298
Title: CAPABLE Care + Connect: Pilot Feasibility of Implementing CAPABLE Into Homebased Primary Care
Brief Title: CAPABLE Care + Connect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); The Rita and Alex Hillman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00471865
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Social Isolation in Older Adults; Social Isolation or Loneliness; Social Isolation; Quality of Life; Disability Physical; Homebound Persons
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: The investigators will have a standard of care group and an intervention group. The intervention group will receive the CAPABLE intervention, and the standard of care group is designed to look at long term outcomes of JHOME patients who did not enroll in CAPABLE compared to those who did.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open-Label Pilot (Experimental): The Open Label Pilot will include testing the CAPABLE Care + Connect intervention on a total of 8. The investigators will recruit and provide CAPABLE to four caregiver-patient dyads (eight participants) and four older adults without caregivers.
  Interventions: Behavioral: CAPABLE Care + Connect - Open Label Pilot
- Pilot- Intervention (Experimental): The investigators will recruit fifteen new partner-patient dyads and fifteen participants without caregivers to receive CAPABLE. That is a total of 45 participants that will receive the CAPABLE intervention
  Interventions: Behavioral: CAPABLE Care + Connect - Pilot
- Standard of Care Group (No Intervention): The standard of care/comparison group will apply for JHOME patients. There are currently around 400-450 patients in JHOME, therefore, our total sample size including both intervention and standard of care group will be up to 450 people.
  It is important to note that the standard of care group is for individuals who did not complete the intervention and is used to evaluate the effectiveness of the intervention itself. Those eligible for the intervention will be included in the study, whereas those ineligible based on intervention screen will be asked about record review. If those ineligible decline record review, those ineligible will be excluded from entire study.

INTERVENTIONS:
Behavioral: CAPABLE Care + Connect - Open Label Pilot — As in CAPABLE, the delivery characteristics of CAPABLE Care + Connect consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW). Adaptations targeting those in JHOME will be made on a per-client basis as part of the open-label pilot. The investigators will further refine and develop the intervention by receiving feedback from the open label pilot participants and CAPABLE clinicians who implemented the pilot to gain those perspectives of the acceptability and feasibility of implementing the CAPABLE Care + Connect intervention. Based on this feedback, the study team will have developed an adapted iteration of the prototype.
  Arms: Open-Label Pilot
Behavioral: CAPABLE Care + Connect - Pilot — As in CAPABLE, the delivery characteristics of CAPABLE Care + Connect consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW). Refinements based on the open label pilot results will be included.
  Arms: Pilot- Intervention

SUMMARY:
In this evaluation scale-up research project, the investigators seek to test an implementation of CAPABLE on the infrastructure of home-based primary care for individuals who may experience social isolation and/or loneliness. These two home-based care programs may improve each other and provide opportunity to further improve quality of life for people living with disabilities and the caregivers. The purpose of this mixed methods study is to adapt and test CAPABLE, an existing evidence-based program, to a new target population with the scalable infrastructure of home-based primary care.

DETAILED DESCRIPTION:
CAPABLE is a home-based, interdisciplinary, goal-directed program that reduces physical disability by working with the person and environment. This program has shown improved performance of activities of daily living (ADL), instrumental activities of daily living (IADL), and depression. Coordinating CAPABLE and Johns Hopkins Home-Based Medicine (JHOME) can help address barriers to health, function, and social connection. Amid limited to no evidence-based strategies to address social isolation and loneliness, this study offers a unique opportunity to address this problem. Because CAPABLE addresses environmental and personal needs to improve the ADL and IADL function of people with disabilities, combining the two programs may better enable people who are homebound to more easily navigate and access the home or beyond. Additionally, this effort will enable the investigators to explore the impact of this combined intervention on social isolation and loneliness.

As in CAPABLE (NA_00031539), the delivery characteristics of CAPABLE Family consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW).

The purpose of this mixed methods study is to adapt and test CAPABLE, an existing evidence-based program, to a new target population with the scalable infrastructure of home-based primary care. The investigators seek to explore if the CAPABLE program increases social connection in homebound older adults, and if the benefits of CAPABLE services improve social connections among socially isolated/lonely homebound older adults.

ELIGIBILITY:
Inclusion Criteria:

* Any patient currently in JHOME
* At risk for or experiencing social isolation as defined by the Lubben Social Network Scale 6 item score less than or equal 12 points or loneliness as defined by the UCLA Loneliness Scale 3 item score of 6 to 9 points
* Cognitive inclusion criteria Montreal Cognitive Assessment (MOCA) >23 as determined by referring JHOME study team member provider
* English speaking (measures are standardized in English)
* Ability to participate in an approximately 45-60 min virtual or in person meeting
* Eligible for CAPABLE
* 50 years or older
* Not hospitalized over night more than 4 times in the last 12 months
* Have some difficulty with any ADL
* Cognitively intact
* Live in Baltimore County or Baltimore City
* Not receiving active cancer treatment
* Interested in participating in CAPABLE Care partners will be included if the care partners provide > 10 hours of care/week

Exclusion Criteria:

* Terminally ill
* live in long term care setting
* receiving active cancer treatment

Standard of Care/Comparison group Inclusion Criteria:

• Any patient currently in JHOME who did not receive the CAPABLE intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Function as assessed by the Katz Index of Independence in Activities of Daily Living Scale | Baseline, 16 weeks
  6 questions, each 1 point for a total score range of 1- 6. A score closer to 6 indicates high patient independence, better outcome.
Change in Function as assessed by Lawton & Brody's assessment of Instrumental Activities of Daily Living Scale (IADL) | Baseline, 16 weeks
  Participants rate their ability to perform daily tasks on a 5-point scale (1 = no difficulty, 2 = a little difficulty, 3 = moderate difficulty, 4 = a lot of difficulty, 5 = unable to do). Score range 8 to 40, higher scores represent greater difficulty performing ADLs, worse outcome.
Change in Pain as assessed by the Brief Pain Inventory Scale (Short Form) | Baseline, 16 weeks
  The Brief Pain Inventory - Short Form is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. For the 10 point scale, 0 indicated no pain and 10 indicates the worst imaginable pain. Score range 0-90, higher score worse outcome.
Change in Function as assessed by the American Community Survey Disability Measure | Baseline, 16 weeks
  This measure is used to identify whether a person is considered to have a disability based on responses to six standardized questions. A person is considered to have a disability if the person answers "Yes" to at least one of the six questions. There is no composite score.
Change in Depression as assessed by the Patient Health Questionnaire Depression Scale (PHQ-8) | Baseline, 16 weeks
  The PHQ-8 contains 8 questions, with a 0-3 scale. A score of 10 or greater is considered major depression, 20 or more is severe major depression. Score range 0-24, higher score worse outcome.
Change in Social Connection as assessed by the Lubben Social Network Scale | Baseline, 16 weeks
  The Lubben Social Network Scale - 12 item version (LSNS-12) includes 12 questions, each scored from 0 to 5 based on the number of social contacts, with total scores ranging from 0 to 60, where lower scores indicate greater social isolation, worse outcome.
Change in Social Connection as assessed by the University of California Los Angeles (UCLA) Loneliness Scale | Baseline, 16 weeks
  The UCLA Loneliness Scale (20-item version) includes 20 questions, each rated on a 1 to 4 scale, with total scores ranging from 20 to 80, where higher scores indicate greater perceived loneliness, worse outcome.
Change in Social Connection as assessed by qualitative questions | Baseline, 16 weeks
  2 open ended questions about social network. Qualitatively look at answers from descriptive perspective
Change in Caregiver Burden as assessed by Zarit Burden Inventory | Baseline, 16 weeks
  The Zarit Burden Interview - 12 item version includes 12 questions, each scored from 0 (never) to 4 (nearly always), for a total score range of 0 to 48, with higher scores indicating greater caregiver burden, worse outcome.
Change in Perceived Change in Function Scale | 16 weeks
  14 questions related to perceived improvement in function. Scale of -2 (gotten much worse) to 2 (improved a lot). The higher the overall score, the greater the improvement, better outcome.
Change in Caregiver Burden as assessed by the Oberest Caregiver Burden Scale | Baseline, 16 weeks
  The Oberst Caregiver Burden Scale includes 15 items rated on a 5-point scale assessing the time and difficulty of caregiving tasks, with total scores ranging from 15 to 75 per subscale and higher scores indicating greater burden.
Change in Caregiver Outcomes as assessed by the Bakas Caregiving Outcomes Scale | Baseline, 16 weeks
  The Bakas Caregiving Outcomes Scale includes 15 items, each rated on a 7-point scale from -3 (changed for the worst) to +3 (changed for the best), with total scores reflecting the caregiver's perceived changes in life due to caregiving. Higher score better.
Change in Pain as assessed by the Brief Pain Inventory (Short Form) | Baseline, 16 weeks
  The Brief Pain Inventory - Short Form is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning on a 10 point scale. 0 = no pain and 10 indicates the worst imaginable pain. Higher score worse outcome.
Change in Pain as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form | Baseline, 16 weeks
  The PROMIS Pain Interference Short Form includes 6 questions, each rated on a 5-point scale, with raw scores summed and converted to a T-score, where higher scores indicate greater interference from pain in daily activities.

SECONDARY OUTCOMES:
JHOME Health System Effects- Number Urgent Visits | 6 months prior to program, 16 weeks
  Frequency (number) of urgent visits
JHOME Health System Effects- Number Emergency Room Visits | 6 months prior to program, 16 weeks
  Frequency (number) of emergency room visits
JHOME Health System Effects - Nursing Home Placement | 16 weeks
  Yes/No to being placed in nursing home
JHOME Health System Effects- Number of Medications | 6 months prior to program, 16 weeks
  Number of medications prescribed

OTHER OUTCOMES:
JHOME Health System Effects- Number Routine Care Visits | 6 months prior to program, 16 weeks
  Frequency (number) of routine care visits

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cudjoe, MD, MPH, MA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No